CLINICAL TRIAL: NCT04502667
Title: Efficacy of Vitamin D Treatment in Pediatric Patients Hospitalized by COVID-19: Open Controlled Clinical Trial
Brief Title: Efficacy of Vitamin D Treatment in Pediatric Patients Hospitalized by COVID-19
Acronym: COVID-19
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Coordinación de Investigación en Salud, Mexico (Other Government)
Collaborators: Hospital Infantil de Mexico Federico Gomez (Other); Hospital General de México Dr. Eduardo Liceaga (Other Government)
Responsible Party: Principal Investigator, Jessie Nallelly Zurita Cruz, principal investigator, Coordinación de Investigación en Salud, Mexico
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R-2020-3603-020
Record Dates: First submitted 2020-08-04; First posted 2020-08-06 (Actual); Last update posted 2022-04-08 (Actual); Status verified 2022-04

CONDITIONS: Covid19; Vitamin D; Children, Only
MeSH Terms: conditions — COVID-19 | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Intervention Model Description: Open controlled clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- cholecalciferol (Vitamin D) (Experimental): Children under 12 months they will be given 1000U and in children over 12 months they will be given 2000U every 24 hours orally during hospitalization
  Interventions: Drug: Cholecalciferol
- Control (No Intervention): No intervention

INTERVENTIONS:
Drug: Cholecalciferol — 1000U or 2000U every 24 hours orally
  Other Names: vitamin D
  Arms: cholecalciferol (Vitamin D)

SUMMARY:
Open controlled clinical trial. Hospitalized pediatric patients with COVID-19 will be included. Upon admission to hospital serum determination of vitamin D, interleukins, ferritin and Dimer D will be performed. Subsequently, randomization will be performed to identify which group the patient belongs. Adverse effects will be evaluated on a daily basis. Serum levels of interleukin (IL) -2, 6, 7,10, ferritin and dimer-D will be taken at the beginning of hospitalization and on the 7th day after admission. It will be recorded if the patient presents deterioration of the respiratory function that requires endotracheal intubation and / or admission to intensive care and / or if he dies, and at what time of hospitalization does this outcome occur. The study will culminate when the patient is discharged from hospitalization.

DETAILED DESCRIPTION:
Hospitalized pediatric patients with COVID-19 will be included. The diagnosis of COVID-19 performed through RT-PCR. Upon admission to hospital, a serum determination of Vitamin D, interleukins, ferritin and dimer-D will be performed. Subsequently, randomization will be performed to identify which group the patient belongs to. In case of being in the vitamin D group, in children under 12 months they will be given 1000U and in children over 12 months they will be given 2000U every 24 hours orally. Adverse effects will be evaluated on a daily basis. Subsequently, serum levels of interleukin (IL) -2, 6, 7,10, ferritin and dimer-D will be taken on day 7 of admission. It will be recorded if the patient presents deterioration of the respiratory function that requires endotracheal intubation and / or admission to intensive care and / or if he dies, and at what time of hospitalization does this outcome occur. The study will culminate when the patient is discharged from hospitalization. On the day of hospital discharge, a blood sample will be taken to determine vitamin D.

ELIGIBILITY:
Inclusion criteria

1. Age over 1 month and under 17 years
2. Confirmed diagnosis of COVID-19 infection with the results of real-time PCR
3. That they agreed to participate in the study.
4. That the patient tolerates the enteral route

Exclusion criteria

1. Have received vitamin D in the four weeks prior to hospitalization.

Ages: 1 Month to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2020-07-15 (Actual); Primary Completion 2021-03-31 (Actual); Study Completion 2021-09-15 (Actual)

PRIMARY OUTCOMES:
INTERLEUKINS (IL-2,6,7,10) (pg/ml) | 7 days
  Taken on admission of the patient to hospitalization (through venipuncture measured by an in-vitro diagnostic enzyme immunoassay (ELISA) for quantitative determination) and on day 7 of hospitalization.
FERRITIN (ng/ml) | 7 days
  Taken on admission of the patient to hospitalization (through venipuncture measured by an in-vitro diagnostic enzyme immunoassay (ELISA) for quantitative determination) and on day 7 of hospitalization.
DIMER-D | 7 days
  Taken on admission of the patient to hospitalization (through venipuncture measured by an in-vitro diagnostic enzyme immunoassay (ELISA) for quantitative determination) and on day 7 of hospitalization.

SECONDARY OUTCOMES:
Vitamin D (ng/ml) | the beginning and through study completion, an average of 21 days
  determination of 25-hydroxy-Vitamin D in human serum

CONTACTS AND LOCATIONS:
Overall Officials: JESSIE ZURITA-CRUZ, Principal Investigator — Coordinación de Investigación en Salud, Mexico
Locations (1):
- Hospital Centro Medico Nacional Siglo XXI, Mexico City, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zurita-Cruz J, Fonseca-Tenorio J, Villasis-Keever M, Lopez-Alarcon M, Parra-Ortega I, Lopez-Martinez B, Miranda-Novales G. Efficacy and safety of vitamin D supplementation in hospitalized COVID-19 pediatric patients: A randomized controlled trial. Front Pediatr. 2022 Jul 25;10:943529. doi: 10.3389/fped.2022.943529. eCollection 2022. PMID 35958172